CLINICAL TRIAL: NCT00938769
Title: Enhanced Self-Efficacy Training For Informal Cancer Caregivers
Brief Title: Enhanced Self-Efficacy Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00009040; 1P01NR010948-01 (NIH)
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Neoplasms
Keywords: cancer; caregiver; symptom; self management
MeSH Terms: conditions — Neoplasms | interventions — Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-Efficacy Training for Caregivers (Other): The Enhanced Caregiver Training intervention will be delivered to informal caregivers of cancer patients before hospital discharge who are randomly selected to receive this intervention. Subjects in the treatment group will receive an individualized experiential caregiver training in strategies for managing patient's symptoms and in the use of pleasant imagery and muscle relaxation to manage stress.
  Interventions: Other: Self-Efficacy Training for Caregivers
- Comparison Conditions for Caregivers (Other): Subjects randomly selected to participate in the attention control training will receive an informational session about cancer and resources for support.
  Interventions: Other: Comparison Conditions for Caregivers

INTERVENTIONS:
Other: Self-Efficacy Training for Caregivers — The Enhanced Caregiver Training intervention will be delivered to informal caregivers of cancer patients before hospital discharge who are randomly selected to receive this intervention. Subjects in the treatment group will receive an individualized experiential caregiver training in strategies for managing patient's symptoms and in the use of pleasant imagery and muscle relaxation to manage stress.
  2-hour in-person instruction of home care issues for caregivers of patients with cancer.
  Arms: Self-Efficacy Training for Caregivers
Other: Comparison Conditions for Caregivers — Subjects randomly selected to participate in the attention control training will receive an informational session about cancer and resources for caregiving.
  2-hour counseling session for cancer caregivers to locate community support resources
  Arms: Comparison Conditions for Caregivers

SUMMARY:
The goal of this study is to examine the effects of an enhanced caregiver training protocol that not only teaches informal caregivers knowledge and skills for managing patient symptoms, but also provides strategies for managing their own psychological distress. The investigators anticipate this training will increase caregivers' self-efficacy and improve important caregiver outcomes (depression, anxiety, burden, quality of life) and patient outcomes (symptom distress/intensity, depression, anxiety, and quality of life). The study will compare the effects of this protocol to an education control condition that equates for interventionist time and attention.

DETAILED DESCRIPTION:
Symptom management is essential in home caregiving. However, many informal caregivers are not confident of their ability to assist their their loved ones with their cancer symptoms at home. A low level of confidence or self-efficacy may negatively affect a caregiver's psychological well-being which is already vulnerable as a consequence of caregiving. Because of the reciprocal nature in a caregiver-patient dyad, caregiver decline is likely associated with patient decline. Improving caregivers' self-efficacy to manage their loved ones' cancer-related symptoms may mitigate their psychological decline and may positively affect patients' well-being by alleviating their symptom distress. Additionally, training in self-management of stress may promote coping among caregivers as many data show that caregiver stress is overwhelming.

This study will examine the effects of an Enhanced Caregiver Training protocol delivered to informal caregivers of cancer patients before hospital discharge. The primary aim is to test the effects of the training on caregivers' self-efficacy in cancer symptom management and self-efficacy in self-management of stress. The study will also look at the effects of this training on caregiver outcomes (depression, anxiety, quality of life, caregiver stress) and patient outcomes (symptom distress and intensity, depression, anxiety, quality of life). The study will use a treatment and attention-control group. Subjects in the treatment group will receive an individualized experiential caregiver training in strategies for managing patient's symptoms and in the use of pleasant imagery and muscle relaxation to manage stress, whereas subjects in the attention-control group will receive an informational session about cancer and resources for caregiving. Data will be collected before and after the training, and at 2 and 4 weeks after hospital discharge. Descriptive statistics and multivariate analysis including mixed models will be used for data analysis This study could have important implications for the nursing community on how to effectively prepare informal cancer caregivers for home caregiving prior to hospital discharge. The long term goal is to refine and expand the training so that it can be used to teach and support informal caregivers of patients suffering from other chronic illnesses, and to determine the cost-effectiveness of this training.

ELIGIBILITY:
Inclusion Criteria (patients):

* Diagnosis of cancer (liquid or solid tumor);
* Admitted to DUMC's 9100 or 9300 for cancer treatment or related complications;
* 18 years of age or older;
* Able to read, speak and write in English;
* Anticipates being discharged to home;
* Not referred to hospice;
* Will have home care needs after discharge;
* No major cognitive impairment;
* Has caregiver willing to do study training and surveys.

Inclusion Criteria (caregivers):

* 18 years of age or older;
* Able to read, speak and write in English;
* Interacts with, and provides most of the hands-on care to, patient who meets above criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2009-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Self-efficacy in symptom management | One month

SECONDARY OUTCOMES:
Psychological well-being | One month
Management of psychological distress | One month
Quality of Life | One month

CONTACTS AND LOCATIONS:
Overall Officials: James A Tulsky, MD, Principal Investigator — Duke University School of Nursing; Cristina Hendrix, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Hendrix CC, Bailey DE Jr, Steinhauser KE, Olsen MK, Stechuchak KM, Lowman SG, Schwartz AJ, Riedel RF, Keefe FJ, Porter LS, Tulsky JA. Effects of enhanced caregiver training program on cancer caregiver's self-efficacy, preparedness, and psychological well-being. Support Care Cancer. 2016 Jan;24(1):327-336. doi: 10.1007/s00520-015-2797-3. Epub 2015 Jun 12. PMID 26062925